CLINICAL TRIAL: NCT05290467
Title: A Reduced-visit Antenatal Care Model Combined With Online Services for Low-risk Pregnant Women
Brief Title: Reduced-visit Antenatal Care Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking University (Other); Peking University China Center for Health Development Studies (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PUTHOGO2ORCT
Record Dates: First submitted 2021-11-09; First posted 2022-03-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2021-10

CONDITIONS: Antenatal Care; Telehealth Services

STUDY DESIGN:
Intervention Model Description: ANC will be provided by obstetricians, and health education will be provided online by midwives. Obstetricians will schedule appointments for the succeeding contacts/visits of the participants. CSOG-recommended prenatal care services will be provided to both the experimental and control groups, using different delivery strategies. Participants in the control group will be scheduled for 12 routine ANC visits, and those in the experimental group will be scheduled for 9 outpatient visits and additional 3 times of services through an online medical service platform. The obstetricians/midwives will train pregnant women how to monitor and record their weight, heart rate, blood pressure, urinary protein, blood glucose, and fetal movement at home. Message, audio and video chats will be used at online ANC contacts to ensure service quality and accuracy of monitoring the results.
Who Masked: Investigator, Outcomes Assessor
Masking Description: ANC allocation will be concealed from investigators who will enroll and assign the participants. Participants and care providers will not be masked to the allocation because of the nature of the ANC, while the outcome assessors and data statistical analysts will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): ANC will be provided by obstetricians, and health education will be provided online by midwives. Obstetricians will schedule appointments for the succeeding contacts/visits of the participants. CSOG-recommended prenatal care services will be provided to the control group. Participants will be scheduled for 12 routine ANC visits.
- experimental group (Experimental): ANC will be provided by obstetricians, and health education will be provided online by midwives. Obstetricians will schedule appointments for the succeeding contacts/visits of the participants. CSOG-recommended prenatal care services will be provided to the experimental group. Participants will be scheduled for 9 outpatient visits and additional 3 times of services through an online medical service platform. The obstetricians/midwives will train pregnant women how to monitor and record their weight, heart rate, blood pressure, urinary protein, blood glucose, and fetal movement at home. Message, audio and video chats will be used at online ANC contacts to ensure service quality and accuracy of monitoring the results.
  Interventions: Behavioral: Online antenatal care

INTERVENTIONS:
Behavioral: Online antenatal care — ANC will be provided by obstetricians, and health education will be provided online by midwives. Obstetricians will schedule appointments for the succeeding contacts/visits of the participants. CSOG-recommended prenatal care services will be provided to both the experimental and control groups, using different delivery strategies. Participants in the control group will be scheduled for 12 routine ANC visits, and those in the experimental group will be scheduled for 9 outpatient visits and additional 3 times of services through an online medical service platform. The obstetricians/midwives will train pregnant women how to monitor and record their weight, heart rate, blood pressure, urinary protein, blood glucose, and fetal movement at home. Messages, audio and video chats will be used at online ANC contacts to ensure service quality and accuracy of monitoring the results.
  Arms: experimental group

SUMMARY:
Antenatal care (ANC) is a critical measure to reduce maternal and perinatal morbidity and mortality. However, there are issues of too many visits and cumbersome procedures of ANC in many maternity hospitals of China. In the past year, the COVID-19 pandemic has brought huge impacts on the health systems, but also gives a valuable chance to review healthcare delivery strategies. Reduced-visit antenatal care models combined with remote monitoring have been recommended and implemented at most hospitals in China during the pandemic, particularly for low-risk pregnant women. However, due to limited evaluations of the cost-effectiveness, policymakers remain confused on how to appropriately integrate online delivery strategies with routine models to improve ANC quality and efficiency sustainably at scale.

This is a single-blind, randomized controlled trial, conducted among low-risk pregnant women at Peking University Third Hospital in Beijing, to evaluate the effectiveness, acceptability, and cost of a reduced-visit ANC model combined with online monitoring compared to the routine ANC model. Participants will be randomly assigned in a 1:1 ratio to receive 12 routine ANC visits or the new ANC model consist of 9 outpatient visits and three online services with remote monitoring on their weight, heart rate, blood pressure, urinary protein, blood glucose, and fetal movement. CSOG-recommended ANC services will be provided to all participants. According to the study objectives and hypotheses, the primary outcome is adverse maternal and perinatal outcomes for non-inferiority analysis, and the secondary outcomes are acceptability and cost for superiority analysis.

DETAILED DESCRIPTION:
Main project problem Is it possible to develop a reduced-visit antenatal care model for low-risk pregnant women, which is more convenient and lower-cost while has same protection for maternal and fetal health compared with routine care? Goals and objectives This project aims to evaluate the acceptability, cost and effectiveness of a reduced-visit antenatal care model combined with online monitoring for low-risk pregnant women, so as to provide evidence for improving antenatal care delivery strategies.

Methods Design, settings and participants A randomized controlled trial will be conducted at the obstetric outpatient department of a tertiary hospital in Beijing between 2022 and 2024. Pregnant women meeting the following criteria are eligible: at 20-34 years old, at <8 weeks of gestation, being registered and scheduled for antenatal care and delivery at this hospital, and without adverse pregnancy-related or medical conditions prior to registration.

Randomization and blinding Pregnant women who complete the first antenatal examination will be assessed for eligibility and recruited by an obstetric nurse. After informed consent is obtained, participants will be randomly assigned to either experimental or control groups using a computer program by an independent statistician blinded to participants' characteristics and health conditions. Obstetricians and nurses provide assigned antenatal care. The outcome assessors and data statistical analysts will be blinded to antenatal care allocation.

Intervention and control methods Participants in the control group will be scheduled for routine 12 clinic visits for antenatal examinations. Participants in the experimental group will be scheduled for 9 clinic visits and additional 3 times of services provided through an online medical service platform. Home self-monitoring for weight, heart rate, blood pressure, urinary protein, blood glucose, and fetal movement is recommended in experimental group, according to the guideline of the Chinese Society of Obstetrics and Gynecology (CSOG) . Such a combination is generally in line with the WHO and CSOG recommendations. Participants developing any complications during pregnancy will be treated according to the conventional clinical pathway, regardless of their grouping.

Data collection and evaluation Participants will be followed up until delivery. Antenatal care time, type and practices will be recorded in detail. Effectiveness, as the primary outcome, will be evaluated by comparing maternal and perinatal outcomes between the two groups. The health outcomes can be extracted from medical records, including maternal, fetal, and neonatal complications, cesarean delivery, preterm, birthweight, Apgar scores, etc. The secondary outcomes include acceptability and cost of the new antenatal model. Acceptability will be measured by comparing satisfaction with antenatal care and pregnancy-related stress. We will measure pregnant women's expectations with prenatal care at 8 weeks of gestation and measure their satisfaction with prenatal care after each visit/contact, using the Patient Expectations and Satisfaction with Prenatal Care (PESPC) instrument. Pregnancy-related stress will be measured at 12, 26 and 36 weeks of gestation by the Pregnancy Stress Rating Scale (PSRS) which has been well validated and widely used (Chen, 2015). Cost of both routine and reduced-visit antenatal care models will be measured from the perspective of both service providers and pregnant women. For a pregnant woman during whole pregnancy, the cost of providing routine antenatal care is calculated by multiplying the average time spent by clinicians and nurses by their average hourly income, and the cost of obtaining antenatal care is calculated by summing the following items: (a) Direct medical cost; (b) Direct non-medical costs, including transportation expenses, accompanying expenses, accommodation expenses, etc. for obtaining prenatal health care services; (c) Indirect costs, calculated by multiplying the working hours delayed by the participants and their families due to antenatal care throughout pregnancy by their normal average hourly income.

Sample size The sample size can be calculated based on expected effectiveness which is considered as the most important endpoint. Given the estimated composite rate of 15% for maternal and perinatal adverse outcomes, a sample size of 1762 patients (881 in each group) would be required with 5% (two-sided) type I error, 80% power, and 10% attrition using a 5% non-inferiority margin.

Statistical Analysis Both intention-to-treat and per-protocol analyses will be performed to account for participants with protocol violations. Satisfaction with antenatal care, pregnancy-related stress, cost, and health outcomes will be compared by arm using independent t-test or one-way analysis of variance for continuous variables and χ2 test or Fisher's exact test for nominal variables. If appropriate, non-inferiority tests will be used by taking a one-sided test of 2.5%, a non-inferiority value of 5%. Multivariable adjusted analyses will be performed to detect the differences more accurately after adjusting for baseline characteristics.

Cost-effectiveness analysis A cost-effectiveness analysis comparing the two ANC models will be conducted by estimating the incremental cost-effectiveness ratios (ICERs) from the perspective of both providers and pregnant women. ICERs are computed by dividing the incremental costs with the differences between the intervention and control groups in primary and secondary outcomes. A sensitivity analysis will be conducted to assess the sensitivity of the cost-effectiveness results with respect to variations in key parameters, including cost.

Expected results and products By the trial, we expect to evaluate the acceptability, cost and effectiveness of the reduced-visit antenatal care model combined with online monitoring. The model will be widely recommended as an alternative method to delivery antenatal care if meeting expectation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19-34 years, ≤8 weeks of gestation, registered and scheduled for ANC and delivery at Peking University Third Hospital, and documented as low risk.

Exclusion Criteria:

* Includes any of the following pregnancy-related or medical conditions: pregnancies by in vitro fertilization, multifetal gestation, BMI ≥28, diabetes, hypertension disorders, thyroid diseases, circulatory diseases, respiratory diseases, nephropathy, inflammatory bowel disease, hepatopathy, coagulopathies, immunodeficiency conditions, mental health disorders, genetic disorders, >2 pregnancy losses, history of preterm delivery at <37 weeks of gestation or stillbirth, and other conditions judged by obstetricians as high-risk pregnancy.

Ages: 19 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1762 (Estimated)
Dates: Start 2022-03-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
A composite rate of adverse maternal and perinatal outcomes | Health outcomes listed as the primary outcome will be extracted from the medical record within one week after delivery or termination of pregnancy.
  The primary outcome, which will be used to address the effectiveness and safety of the adapted ANC model, is the composite rate of adverse maternal and perinatal outcomes defined as the occurrence of any of the following events: maternal death, loss of pregnancy, stillbirth, neonatal death, maternal severe complications (such as gestational hypertension, preeclampsia/eclampsia, anemia, preterm delivery, indicated and emergency cesarean section, puerperal infection, third- or fourth-degree perineal lacerations, uterine rupture, postpartum hemorrhage, blood transfusion, hysterectomy, stroke, organ failure, and admittance to the ICU), fetal and neonatal severe complications (such as fetal growth restriction, low birth weight, macrosomia, birth trauma, neonatal infection, 5-min Apgar scores <7 points, and referral and admittance to the neonatal ICU), and any other pregnancy-associated complications. Health outcomes will be extracted from medical records after each ANC visit or contact.

SECONDARY OUTCOMES:
Satisfaction with antenatal care | Pregnant women's satisfaction with prenatal care will be measured within one week after delivery or termination of pregnancy by calculating average score of PESPC performed at each ANC visit or contact.
  Expectations and satisfaction with ANC will be measured using the Patient Expectations and Satisfaction with Prenatal Care (PESPC) instrument. The PESPC, developed by Omar and colleagues in 2001, consists of 41 items categorized into two subscales consisting of eight dimensions: personalized care (4 items), complete care (4 items), provider continuity (2 items), and other services (2 items) in the expectation subscale and information (7 items), provider care (6 items), staff interest (6 items), and system characteristics (10 items) in the satisfaction subscale. The response options of each item range from 1 (strongly agree) to 6 (strongly disagree), with no neutral response option. The PESPC was found to be a valid and reliable self-report instrument of ANC quality. Pregnant women's satisfaction with prenatal care will be measured within one week after delivery or termination of pregnancy by calculating average score of PESPC performed at each ANC visit or contact.
Pregnancy-related stress | Pregnancy-related stress will be measured within one week after delivery or termination of pregnancy by calculating average score of PSRS performed at 12, 26, and 36 weeks of gestation.
  Pregnancy-related stress will be measured at 12, 26, and 36 weeks of gestation using the Pregnancy Stress Rating Scale (PSRS), which has been well validated and widely used. The PSRS was initially developed in 1983 and revised and validated in 2015 by Chen et al. The revised PSRS consists of 36 items indicating potentially stressful pregnancy-related events and anticipated events during the labor, delivery, and immediate postpartum periods, which may come from the following: (a) seeking safe passage for mother and child through pregnancy, labor, and delivery, (b) infant care and changing family relationships, (c) maternal role identification, (d) social support seeking, and (e) altered physical appearance and function. The revised PSRS is found to be psychometrically sound in assessing prenatal stress in Chinese women.
Antenatal care cost | ANC costs will be measured from the perspectives of both service providers and pregnant women after delivery or termination of pregnancy.
  ANC costs will be measured from the perspectives of both service providers and pregnant women after each ANC visit or contact. For a pregnant woman during the entire pregnancy, the cost of providing routine ANC is calculated by multiplying the average time spent by clinicians and nurses with their average hourly income, and the cost of obtaining ANC is calculated by summing the following items: (a) Direct medical cost; (b) Direct non-medical costs, including transportation expenses, accompanying expenses, accommodation expenses, etc. for obtaining prenatal health care services; (c) Indirect costs, calculated by multiplying the working hours delayed by participants and their families due to antenatal care throughout pregnancy by their normal average hourly income. The ANC provision and utilization costing forms will be initially developed by our research team and then revised by an expert panel consisting of obstetricians, midwives, nurses, health economists, and questionnaire experts.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Requested data for public purpose or research transparency will be provided via the corresponding author after 36 months following trial completion.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Requested data for public purpose or research transparency will be provided via the corresponding author after 36 months following trial completion.
Access Criteria: Requested data for public purpose or research transparency will be provided via the corresponding author. The e-mail address is weiyuanbysy@163.com.

REFERENCES:
- [Derived] Shi H, Wang Y, Dang B, Li D, Ma S, Wang X, Li Z, Hao W, Li C, Jiang Y, Yuan P, Chen L, Gong X, Wang Y, Wu X, Zhao Y, Wei Y. Reduced-visit antenatal care model combined with telemedicine for low-risk pregnant women: protocol for a randomised controlled trial. BMJ Open. 2023 Jul 21;13(7):e067110. doi: 10.1136/bmjopen-2022-067110. PMID 37479506